CLINICAL TRIAL: NCT02978521
Title: Effect of a Pulmonary Rehabilitation Program on Skeletal Muscle Mass, Pulmonary Function, Inflammatory Response and Overall Survival on Patients Diagnosed With Non-small-cell Advanced Cancer
Brief Title: Pulmonary Rehabilitation in Advanced Non-small Cell Lung Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Principal Investigator, Head of the Thoracic Oncology Unit, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 016/028/ICI
Record Dates: First submitted 2016-11-18; First posted 2016-12-01 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Rehabilitation; Sarcopenia; Quality of Life
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): Patients in the IG will be scheduled to receive Pulmonary Rehabilitation:
  12 sessions (60 minutes approximately) over a period of 4-6 weeks (2-3 session/week). Sessions will progress as patients tolerance to exercise and will include breathing techniques, resistance training on ergometer and treadmill.
  Interventions: Other: Pulmonary rehabilitation
- Control Group (No Intervention): CG will receive information and recommendations on physical activity

INTERVENTIONS:
Other: Pulmonary rehabilitation — Session 1: ventilatory pattern training Session 2,3: ventilatory pattern + respiratory training with incentive spirometer Session 4-6: Sessions 1-3 training continues + training with Positive expiratory pressure device (Threshold PEP) and breathing trainer Threshold IMT) Sessions 7-9: Continue respiratory training + resistance training with RECK MOTOmed2 ergometer at a 30% intensity until 60% is achieved Session 10-12: Continue with previous training + treadmill training
  Arms: Intervention Group

SUMMARY:
Lung cancer (LC) is usually diagnosed in advanced stages and continues to be the leading cause of cancer related deaths worldwide. Cancer cachexia are frequent among patients with LC affecting up to 80% of patients with advanced stage disease, and it has been related with higher risk of complications, length of hospital stay, and worst overall survival. During cancer cachexia, both muscle and fat mass can be wasted, however, the loss of muscle mass has been associated to higher treatment related toxicity, loss of functional status, shorter progression free survival and overall survival in different types of cancer under various treatments. Hence, preservation of muscle mass and function should be an important focus of the multidisciplinary treatment of patients with LC.

Pulmonary rehabilitation (PR) has been known to improve pulmonary function, reduce fatigue and improve exercise tolerance in patients with LC undergoing curative surgery. However, few studies have focused on the efficacy of PR on patients with advanced cancer undergoing palliative care with chemotherapy or targeted therapies.

DETAILED DESCRIPTION:
The main objective of this study is to determine the effects of a pulmonary rehabilitation program on the pulmonary function and muscle mass. Moreover, the effects on exercise tolerance, inflammatory response, quality of live and overall survival will be explored.

Patients will be randomized into intervention group (IG) or control group (CG). Patients in the IG will be scheduled to receive 12 sessions of PR over a period of 4-6 weeks (2-3 session/week). CG will receive information and recommendations on physical activity. Both groups will receive nutritional assessment and intervention as needed.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of advanced non-small-cell lung cancer
* Good performance status (ECOG 0-1)
* Life expectancy >12 weeks
* Eligible to receive treatment with chemotherapy or tyrosinkinase inhibitors
* Recent electrocardiogram without evidence of arrythmia

Exclusion Criteria:

* Symptomatic brain metastasis
* Uncontrolled pain (Visual Analog Scale >5)
* Uncontrolled hypertension (>140/100mmHg)
* Practice of regular moderate to intense physical activity at least 3 day/week
* Not residents of Mexico City or unable to attend to therapy sessions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2016-08-05 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function | After 12 sessions (6 weeks)
  Pulmonary function Maximal expiratory and inspiratory pressure units: cm H2O (measured with Jaeger spirometer)

SECONDARY OUTCOMES:
Muscle mass | After 12 sessions (6 weeks)
  Muscle mass measured by body composition analysis of CT images using lumbar vertebra 3 (L3)
Inflammatory response | After 12 sessions (6 weeks)
  Quantification of: Interleukin (IL)-8, IL-1β, IL-6, IL-10, IL-12 and tumor necrosis factor (TNF) (Human Inflammatory Cytokine Kit Becton, Dickinson and Company (BD)™ Cytometric Bead Array) Units: pg/ml
Exercise tolerance | After 12 sessions (6 weeks)
  6 minute walk test
Quality of Life in lung cancer | the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire is applied before and after a follow-up after 12 sessions (6 weeks).
  To determine the Quality of Life (QoL) of patients with lung cancer and its association with rehabilitation.
  Application of the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire, the EORTC QLQ-C30. It is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. It ranges in score from 0 to 100. A high scale score represents a higher response level.
Lung Cancer Quality of Life | After 12 sessions (6 weeks)
  Application of the "european organization for research and treatment of cancer quality of life questionnaire (QLQ)LC-13"
Anxiety and Depression | After 12 sessions (6 weeks)
  Hospital Anxiety and Depression Scale (HADS

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, Study Director — Head of Thoracic Oncology Unit
Locations (1):
- Instituto Nacional de Cancerología, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruera E. ABC of palliative care. Anorexia, cachexia, and nutrition. BMJ. 1997 Nov 8;315(7117):1219-22. doi: 10.1136/bmj.315.7117.1219. No abstract available. PMID 9393230
- [Background] Argiles JM, Alvarez B, Lopez-Soriano FJ. The metabolic basis of cancer cachexia. Med Res Rev. 1997 Sep;17(5):477-98. doi: 10.1002/(sici)1098-1128(199709)17:53.0.co;2-r. No abstract available. PMID 9276862
- [Background] Blum D, Omlin A, Baracos VE, Solheim TS, Tan BH, Stone P, Kaasa S, Fearon K, Strasser F; European Palliative Care Research Collaborative. Cancer cachexia: a systematic literature review of items and domains associated with involuntary weight loss in cancer. Crit Rev Oncol Hematol. 2011 Oct;80(1):114-44. doi: 10.1016/j.critrevonc.2010.10.004. Epub 2011 Jan 8. PMID 21216616
- [Background] Rhee CM, Kalantar-Zadeh K. Resistance exercise: an effective strategy to reverse muscle wasting in hemodialysis patients? J Cachexia Sarcopenia Muscle. 2014 Sep;5(3):177-80. doi: 10.1007/s13539-014-0160-z. Epub 2014 Aug 28. PMID 25163460
- [Background] Ozalevli S, Ilgin D, Kul Karaali H, Bulac S, Akkoclu A. The effect of in-patient chest physiotherapy in lung cancer patients. Support Care Cancer. 2010 Mar;18(3):351-8. doi: 10.1007/s00520-009-0659-6. Epub 2009 May 28. PMID 19471973
- [Background] Tarumi S, Yokomise H, Gotoh M, Kasai Y, Matsuura N, Chang SS, Go T. Pulmonary rehabilitation during induction chemoradiotherapy for lung cancer improves pulmonary function. J Thorac Cardiovasc Surg. 2015 Feb;149(2):569-73. doi: 10.1016/j.jtcvs.2014.09.123. Epub 2014 Oct 5. PMID 25451483
- [Background] Mourtzakis M, Prado CM, Lieffers JR, Reiman T, McCargar LJ, Baracos VE. A practical and precise approach to quantification of body composition in cancer patients using computed tomography images acquired during routine care. Appl Physiol Nutr Metab. 2008 Oct;33(5):997-1006. doi: 10.1139/H08-075. PMID 18923576
- [Background] Prado CM, Lieffers JR, McCargar LJ, Reiman T, Sawyer MB, Martin L, Baracos VE. Prevalence and clinical implications of sarcopenic obesity in patients with solid tumours of the respiratory and gastrointestinal tracts: a population-based study. Lancet Oncol. 2008 Jul;9(7):629-35. doi: 10.1016/S1470-2045(08)70153-0. Epub 2008 Jun 6. PMID 18539529
- [Background] Degner LF, Sloan JA. Symptom distress in newly diagnosed ambulatory cancer patients and as a predictor of survival in lung cancer. J Pain Symptom Manage. 1995 Aug;10(6):423-31. doi: 10.1016/0885-3924(95)00056-5. PMID 7561224
- [Background] Stigt JA, Uil SM, van Riesen SJ, Simons FJ, Denekamp M, Shahin GM, Groen HJ. A randomized controlled trial of postthoracotomy pulmonary rehabilitation in patients with resectable lung cancer. J Thorac Oncol. 2013 Feb;8(2):214-21. doi: 10.1097/JTO.0b013e318279d52a. PMID 23238118
- [Background] Rivas-Perez H, Nana-Sinkam P. Integrating pulmonary rehabilitation into the multidisciplinary management of lung cancer: a review. Respir Med. 2015 Apr;109(4):437-42. doi: 10.1016/j.rmed.2015.01.001. Epub 2015 Jan 22. PMID 25641113
- [Background] Jastrzebski D, Maksymiak M, Kostorz S, Bezubka B, Osmanska I, Mlynczak T, Rutkowska A, Baczek Z, Ziora D, Kozielski J. Pulmonary Rehabilitation in Advanced Lung Cancer Patients During Chemotherapy. Adv Exp Med Biol. 2015;861:57-64. doi: 10.1007/5584_2015_134. PMID 26017725
- [Background] Henke CC, Cabri J, Fricke L, Pankow W, Kandilakis G, Feyer PC, de Wit M. Strength and endurance training in the treatment of lung cancer patients in stages IIIA/IIIB/IV. Support Care Cancer. 2014 Jan;22(1):95-101. doi: 10.1007/s00520-013-1925-1. Epub 2013 Sep 1. PMID 23995813
- [Background] Hwang CL, Yu CJ, Shih JY, Yang PC, Wu YT. Effects of exercise training on exercise capacity in patients with non-small cell lung cancer receiving targeted therapy. Support Care Cancer. 2012 Dec;20(12):3169-77. doi: 10.1007/s00520-012-1452-5. Epub 2012 Apr 14. PMID 22526147